CLINICAL TRIAL: NCT02568683
Title: A Phase 1b-2, Open-Label, Dose Escalation and Expansion Study Evaluating the Safety and Efficacy of Entospletinib (ENTO [GS-9973]) Combined With Vincristine (VCR) in Adult Subjects With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Safety and Efficacy of Entospletinib (ENTO [GS-9973]) Combined With Vincristine (VCR) in Adult Participants With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (NHL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-1562; 2015-002731-17 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: DLBCL; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: ENTO (Experimental): Participants will be enrolled sequentially in a 3 + 3 dose escalation design to receive escalating dose of ENTO+VCR at dose levels 1 to 4 with the objective of defining the maximum tolerated dose (MTD) or recommended dose for the dose expansion stage. Following the determination of the MTD of the dose levels 1 to 4 (or concurrently with the opening of dose level 4), the safety of administering ENTO with VCR when administered as a 4-day prolonged continuous infusion may be evaluated in the continuous infusion dose escalation level (dose level C1) with the objective of investigating the schedule of dosing ENTO when administered with VCR as a continuous infusion.
  Interventions: Drug: Entospletinib; Drug: Vincristine
- Dose Expansion: VCR+ENTO (Cohort A) (Experimental): Based on the tolerability, safety, and efficacy data from the dose escalation phase, participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) may receive VCR+ENTO.
  Interventions: Drug: Entospletinib; Drug: Vincristine
- Dose Expansion: VCR+ENTO (Cohort B) (Experimental): Based on the tolerability, safety, and efficacy data from the dose escalation phase, participants with relapsed or refractory B-cell NHL (non-DLBCL) may receive VCR+ENTO.
  Interventions: Drug: Entospletinib; Drug: Vincristine

INTERVENTIONS:
Drug: Entospletinib — ENTO spray dried dispersion tablets administered orally twice daily while in a fasted state
  Other Names: GS-9973; ENTO
Drug: Vincristine — VCR administered intravenously
  Other Names: VCR

SUMMARY:
The primary objective of this study is to evaluate the safety of ENTO with VCR in participants with relapsed or refractory B-cell NHL.

ELIGIBILITY:
Key Inclusion Criteria:

* Measurable disease by computed tomograph (CT)/ and/or positron-emission tomography CT (PET-CT)
* A) Dose Escalation Stage: Confirmed diagnosis of relapsed or refractory B-Cell NHL treated with prior treatment for lymphoid malignancy comprising of at least 1 regimen containing a therapeutic anti-CD20 antibody (eg, rituximab, ofatumumab, GA-101) and at least 2 prior combination chemotherapy regimens (or autologous stem cell transplant) , or treated with 1 prior combination chemotherapy regimen in patients without an approved second-line therapy option, requiring treatment in the opinion of the treating physician
* B) Dose Expansion Cohorts:

  * Expansion Cohort A: Diagnosis of relapsed or refractory DLBCL treated with prior treatment for lymphoid malignancy comprising of at least 1 regimen containing a therapeutic anti-CD20 antibody (eg, rituximab, ofatumumab, GA-101) and at least 2 prior combination chemotherapy regimens or autologous stem cell transplant, or treated with 1 prior combination chemotherapy regimen in patients without an approved second-line therapy option, requiring treatment in the opinion of the treating physician
  * Expansion Cohort B: Diagnosis of relapsed or refractory B-cell NHL (other than DLBCL) treated with prior treatment for lymphoid malignancy comprising of at least 1 regimen containing a therapeutic anti-CD20 antibody (eg, rituximab, ofatumumab, GA-101) and at least 2 prior combination chemotherapy regimens or autologous stem cell transplant, or treated with 1 prior combination chemotherapy regimen in patients without an approved second-line therapy option, requiring treatment in the opinion of the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky performance status ≥ 70
* Required screening laboratory data (within 2 weeks prior to administration of study drug) as defined in study protocol.
* Adequate organ function defined by the screening laboratory inclusion and Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram (ECHO) or multigated acquisition (MUGA)
* Discontinuation of all therapy (including radiotherapy, chemotherapy, tyrosine kinase inhibitors (TKIs), immunotherapy, or investigational therapy for the treatment of cancer at least 2 weeks prior to the initiation of study therapy
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before enrollment, with the exception of alopecia (any grade permitted)
* For female individuals of childbearing potential, willingness to use a protocol-recommended method of contraception from the Screening visit throughout the study and 30 days from the last dose of ENTO or VCR, whichever is later.
* For male individuals having intercourse with females of childbearing potential, willingness to abstain from heterosexual intercourse or use a protocol-recommended method of contraception from the start of study drug throughout the study treatment period and for 90 days following the last dose of ENTO or VCR, whichever is later and to refrain from sperm donation from the start of the study drug throughout the study treatment period and for 90 days following the last dose of ENTO or VCR, whichever is later.
* In the judgment of the investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the individual's NHL
* Willingness to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions
* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures

Key Exclusion Criteria:

* Diagnosis of Primary Mediastinal Large B-cell Lymphoma
* A life threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the individual's safety or interfere with the absorption or metabolism of ENTO
* Active or symptomatic central nervous system (CNS) disease or epidural involvement
* Uncontrolled intercurrent illness including, but not limited to, unstable angina pectoris or psychiatric illness/social situations that would limit compliance with study requirements
* Current/ongoing Neuropathy (sensory or motor) Grade > 1 or any history of Grade ≥ 3 neuropathy with prior VCR or chemotherapy exposure (documentation by history is adequate to exclude)
* Contraindication to receive VCR or any planned protocol-specified chemotherapy
* Eligible for autologous stem cell transplant
* History of myelodysplastic syndrome, allogeneic stem cell or solid organ transplantation
* History of any other prior lymphoid malignancy other than the registrational histology or any other non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥ 1 year prior to the start of study drug, or any other cancer that has been in complete remission without treatment for ≥ 5 years prior to enrollment
* Known hypersensitivity or intolerance to any of the active substances or excipients in the formulations for ENTO
* Evidence of uncontrolled systemic bacterial, fungal, or viral infection at the start of study drug
* Ongoing drug-induced liver injury, chronic active Hepatitis C Virus (HCV), chronic active Hepatitis B Virus (HBV), human immunodeficiency virus (HIV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension
* Current therapy with proton pump inhibitors
* Pregnancy or breastfeeding
* Ongoing active pneumonitis
* Prior treatment with a spleen tyrosine kinase (SYK) inhibitor

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (2):
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Medical University of South Carolina, Charleston, South Carolina
- France (5):
  - Groupe Hospitalier du Haut Leveque, Pessac, Aquitaine
  - Centre Hospitalier Régional Universitaire de Lille (CHRU de Lille), Lille, Hauts-de-France
  - Institut Paoli Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire de Dijon Hôpital du Bocage, Dijon
  - Centre Hospital Lyon Sud, Pierre-Bénite

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and France. The first participant was screened on 11 February 2016. The last study visit occurred on 22 June 2017.
Pre-assignment Details: 13 participants were screened.
Groups:
- ENTO 200 mg: Participants received entospletinib (ENTO) 200 mg tablet twice daily + vincristine (VCR) 1.0 mg/m^2 administered via intravenous infusion every 14 days; up to 24 weeks.
- ENTO 400 mg: Participants received ENTO 400 mg tablet twice daily + VCR 1.0 mg/m^2 administered via intravenous infusion every 14 days; up to 8 weeks.
Period: Overall Study
Arm/Group | ENTO 200 mg | ENTO 400 mg
Started | 6 | 4
Completed | 0 | 0
Not Completed | 6 | 4
Not completed — Death | 0 | 2
Not completed — Withdrew Consent | 1 | 0
Not completed — Study Terminated By Sponsor | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who received at least 1 dose of ENTO.
Groups:
- ENTO 200 mg: Participants received ENTO 200 mg tablet twice daily + VCR 1.0 mg/m^2 administered via intravenous infusion every 14 days; up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | ENTO 200 mg | ENTO 400 mg | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13.6) | 69 (8.1) | 65 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4 | 1 | 5
  Race: Not Permitted | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 4 | 1 | 5
  Ethnicity: Not Permitted | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Laboratory (Lab) Abnormalities Defined as Dose Limiting Toxicities (DLTs) in Participants With Relapsed or Refractory B-cell NHL: Dose Escalation Stage
Description: Occurrence of any of the following toxicities during Cycle 1 was considered DLT if judged by the Investigator to be possibly, probably, or definitely related to the administration of any drug in the treatment regimen:
  * Grade 4 (or higher) non-hematologic toxicity
  * Grade 3 non-hematologic toxicity lasting ≥ 7 days despite optimal supportive care
    * Note: Grade 3 or higher neuropathy was considered DLT if occurring during Cycle 1 regardless of duration.
  * Any Grade 3 non-hematologic laboratory value if:
    * Medical intervention was required to treat the patient, or
    * Abnormality led to hospitalization, or
    * Abnormality persisted for > 1 week
  * Grade 4 Neutropenia (absolute neutrophil count [ANC] < 500 /μL) persisting for > 14 days or associated with febrile neutropenia
  * Grade 4 thrombocytopenia (platelets < 25,000 cells/μL) persisting for > 14 days (or > 25,000 cells/μL, but requiring prophylactic platelet transfusion to maintain this level)
Time Frame: Cycle 1 (28-day cycle)
Population: DLT Analysis Set included participants in the Full Analysis Set (included all participants who received at least 1 dose of ENTO) who received 37 of 56 Cycle 1 doses of ENTO and completed the full Cycle 1 dose of VCR or who experienced a DLT during the DLT assessment window.
Measure: Count of Participants; unit: Participants
Arm/Group | ENTO 200 mg | ENTO 400 mg
Number analyzed (Participants) | 6 | 3
Participants | 0 | 2

2. Secondary Outcome: Number of Participants With AEs and Lab Abnormalities Not Defined as DLTs in Participants With Relapsed or Refractory B-cell NHL: Dose Escalation Stage
Description: The number of participants with AEs and lab abnormalities not defined as DLTs in participants in the dose escalation stage with relapsed or refractory B-cell NHL are presented.
Time Frame: Cycle 1 (28-day cycle)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | ENTO 200 mg | ENTO 400 mg
Number analyzed (Participants) | 6 | 4
Participants
  AEs not defined as DLTs | 6 | 4
  Lab abnormalities not defined as DLTs | 5 | 4

3. Secondary Outcome: Duration of Exposure to ENTO
Time Frame: Baseline to end of study (maximum: 24 weeks)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | ENTO 200 mg | ENTO 400 mg
Number analyzed (Participants) | 6 | 4
weeks | 17.7 (6.09) | 4.3 (2.68)

4. Secondary Outcome: Number of VCR Doses
Time Frame: Baseline to end of study (maximum: 24 weeks)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | ENTO 200 mg | ENTO 400 mg
Number analyzed (Participants) | 6 | 4
doses | 8.7 (3.27) | 2.3 (1.50)

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 200 mg ENTO = 24 weeks; 400 mg ENTO = 8 weeks)
Description: Full Analysis Set included all participants who received at least 1 dose of ENTO.
Arm/Group | ENTO 200 mg | ENTO 400 mg
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 200 mg (N=6) | ENTO 400 mg (N=4)
Pyrexia (General disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 200 mg (N=6) | ENTO 400 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Feeling drunk (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0
Sepsis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Because the study was terminated after enrolling only 10 participants, the dose expansion stage and the planned efficacy analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years